CLINICAL TRIAL: NCT02701218
Title: Comparison of the Treatment Outcomes of Posterior Canal Benign Paroxysmal Positional Vertigo (BPPV) With Canalith Repositioning Procedure (CRP): Single Versus Multiple Cycles
Brief Title: BPPV With CRP: Single Versus Multiple Cycles
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chiang Mai University (Other)
Responsible Party: Principal Investigator, Suwicha Isaradisaikul Kaewsiri, Principal Investigator, Clinical Professor, Chiang Mai University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ENT-2558-03601
Record Dates: First submitted 2016-02-18; First posted 2016-03-08 (Estimated); Last update posted 2019-07-31 (Actual); Status verified 2019-07

CONDITIONS: Benign Paroxysmal Positional Vertigo (BPPV)
Keywords: Canalith repositioning procedure (CRP); BPPV
MeSH Terms: conditions — Benign Paroxysmal Positional Vertigo

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Single cycle (Experimental): single cycle of canalith repositioning procedure
  Interventions: Procedure: Canalith repositioning procedure
- multiple cycles of CRP (Experimental): multiple cycles of canalith repositioning procedure CRP will be stopped if 1) no nystagmus and vertigo in all positions 2) complications exited 3) stable nystagmus in the 2 last cycles
  Interventions: Procedure: Canalith repositioning procedure

INTERVENTIONS:
Procedure: Canalith repositioning procedure — Canalith repositioning procedure; single or multiple cycles
  Other Names: Epley's maneuver

SUMMARY:
Unilateral posterior canal benign paroxysmal positional vertigo (BPPV) cases will be randomized to treat with single or multiple cycles of canalith repositioning procedure.The treatment outcomes will be assessed at 7th and 28th days.

DETAILED DESCRIPTION:
Patients present with brief episodes of vertigo will be evaluated by Dix-Hallpike test. Cases with positive Dix-Hallpike test, unilateral, posterior canal, will be randomized with block of four. Either single or multiple cycles of canalith repositioning procedure will be performed. Four treatment outcomes will be blindly assessed at 7 and 28 days.

ELIGIBILITY:
Inclusion Criteria:

1. Recurrent episodes of vertigo
2. 15 years of age or older
3. Positive Dix-Hallpike test: unilateral, posterior canal

Exclusion Criteria:

1. Received vestibular suppressant within 6 hours
2. With other diseases or conditions cause of vertigo or central nervous system disease
3. With diseases or conditions contraindicate for Dix-Hallpike test or CRP eg: cervical spine disease, back/ neck stiffness, retinal detachment
4. Positive Dix-Hallpike test: bilateral, other canals
5. Complications from CRP eg: nausea, vomiting, canalith jam
6. Cannot read the questionaire

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2016-02 (Actual); Primary Completion 2019-03 (Actual); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Dix-Hallpike test (DHT) | At 7th day
  percentage of negative DHT between single and multiple cycles

SECONDARY OUTCOMES:
Dizziness handicap inventory (DHI) | compare to the first visit at 7th between single and multiple cycles
  total score in the questionaire
Dizziness handicap inventory (DHI) | compare to the first visit at 28th day between single and multiple cycles
  total score in the questionaire
Subjective symptoms | Improvement of the symptoms compare to the first visit at 7th day between single and multiple cycles
  Asking the patient's symptom: Improve, same, worse
Subjective symptoms | Improvement of the symptoms compare to the first visit at 28th day between single and multiple cycles
  Asking the patient's symptom: Improve, same, worse
Loss of balance | compare to the first visit at 7th between single and multiple cycles
  5 levels Level 1: Able to continue daily activities without any helps. Level 2: Able to continue daily activities without any helps except complicated activities such as riding a bicycle, walking on counterpoise or scaffolding.
  Level 3: Not able to continue daily activities without help excepts simple activities such as self-care, housework, walking, or being a passenger in a vehicle Level 4: Not able to continue daily activities alone without help except self-care Level 5 Not able to continue daily activities alone without help except self-care without ambulation. Need to stay only in a house or a living place.
  (From: The Royal college of Otolaryngologists head and neck surgeons of Thailand, and social security office of thailand)
Loss of balance | compare to the first visit at 28th day between single and multiple cycles
  5 levels Level 1: Able to continue daily activities without any helps. Level 2: Able to continue daily activities without any helps except complicated activities such as riding a bicycle, walking on counterpoise or scaffolding.
  Level 3: Not able to continue daily activities without help excepts simple activities such as self-care, housework, walking, or being a passenger in a vehicle Level 4: Not able to continue daily activities alone without help except self-care Level 5 Not able to continue daily activities alone without help except self-care without ambulation. Need to stay only in a house or a living place.
  (From: The Royal college of Otolaryngologists head and neck surgeons of Thailand, and social security office of thailand)
Dix-Hallpike test (DHT) | At 28th day
  percentage of negative DHT between single and multiple cycles

CONTACTS AND LOCATIONS:
Overall Officials: Suwicha I Kaewsiri, MD, Principal Investigator — Department of Otolaryngology
Locations (1):
- Department of Otolaryngology Faculty of Medicine, Chiang Mai University 110 Intawaroros Road, Sriphum, Chiang Mai, Thailand

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Bhattacharyya N, Baugh RF, Orvidas L, Barrs D, Bronston LJ, Cass S, Chalian AA, Desmond AL, Earll JM, Fife TD, Fuller DC, Judge JO, Mann NR, Rosenfeld RM, Schuring LT, Steiner RW, Whitney SL, Haidari J; American Academy of Otolaryngology-Head and Neck Surgery Foundation. Clinical practice guideline: benign paroxysmal positional vertigo. Otolaryngol Head Neck Surg. 2008 Nov;139(5 Suppl 4):S47-81. doi: 10.1016/j.otohns.2008.08.022. PMID 18973840
- [Derived] Isaradisaikul SK, Chowsilpa S, Hanprasertpong C, Rithirangsriroj T. Single Cycle Versus Multiple Cycles of Canalith Repositioning Procedure for Treatment of Posterior Canal Benign Paroxysmal Positional Vertigo: A Randomized Controlled Trial. Otol Neurotol. 2021 Jan;42(1):121-128. doi: 10.1097/MAO.0000000000002894. PMID 32947492
- Available data/document: Study Protocol: ENT-2558-03601 — http://ros.med.cmu.ac.th/Security/SignIn.aspx — Research administration section website